CLINICAL TRIAL: NCT04010409
Title: Mindreading in Adults With Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201809069RINA
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD Group: Autism spectrum disorder participants, no intervention
  Interventions: Other: no intervention
- TD Group: Typically developmental controls,no intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to investigate the ability of reading emotions by the Eyes task in adults with ASD, and examine the gazing pattern and frontal activation during the task. We plan to recruit 50 adults with ASD and 50 typically-developing adults. Eye-tracking and frontal activation (measured by functional near-infrared spectroscopy) will be examined during the Eyes task.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a clinical syndrome characterized by mindreading deficits, or Theory of Mind deficits. The Reading the Mind in the Eyes task (abbreviated as the Eyes task) was developed to assess the mindreading deficits as a hallmark of social deficits of ASD. This study aims to investigate the ability of reading emotions by the Eyes task in adults with ASD, and examine the gazing pattern and frontal activation during the task. We plan to recruit 50 adults with ASD and 50 typically-developing adults. All the participants will complete clinical measures and the Eyes task. Eye-tracking and frontal activation (measured by functional near-infrared spectroscopy) will be examined during the Eyes task.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged between 20 and 50 years who had a diagnosis of ASD based on DSM-5.
* Had a full-scale IQ > 70 on WAIS-IV.

Exclusion Criteria:

* A history of major mental illness (e.g., bipolar affective disorder, schizophrenia) or neurological diseases.
* Visual impairment and that would preclude participation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The 30 adults with ASD will be recruited from Adult ASD clinics in Department of Psychiatry, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
eye tracking indicators | 30 min
  eye tracking indicators

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ling Chien, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chien YL, Tseng YL, Tsai WC, Chiu YN. Assessing Frontal Lobe Function on Verbal Fluency and Emotion Recall in Autism Spectrum Disorder by fNIRS. J Autism Dev Disord. 2025 May;55(5):1648-1659. doi: 10.1007/s10803-024-06306-5. Epub 2024 Apr 18. PMID 38635133